CLINICAL TRIAL: NCT01389609
Title: Phase 1, Open-Label, Randomized, Single-Dose, 3-Way Crossover Study Assessing Bioequivalence Of Doxazosin 4 Mg Orally-Disintegrating Tablet With Or Without Water To Doxazosin 4 Mg Japanese Marketed Immediate Release Tablet Under Fasted Condition
Brief Title: Bioequivalence Study of Doxazosin 4 Mg Orally-Disintegrating Tablet With Or Without Water To Doxazosin 4 Mg Japanese Marketed Immediate Release Tablet Under Fasted Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A0351069
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Bioequivalence; Orally-disintegrating Tablet
MeSH Terms: conditions — Hypertension | interventions — Doxazosin; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Doxazosin 4 mg Japanese marketed IR tablet as a single oral dose under fasted conditions
  Interventions: Drug: Doxazosin 4 mg Japanese marketed IR tablet
- B (Experimental): Doxazosin 4 mg ODT with water as a single oral dose under fasted conditions
  Interventions: Drug: Doxazosin 4 mg ODT with water
- C (Experimental): Doxazosin 4 mg ODT without water as a single oral dose under fasted conditions
  Interventions: Drug: Doxazosin 4 mg ODT without water

INTERVENTIONS:
Drug: Doxazosin 4 mg Japanese marketed IR tablet — Immediate release tablet, 4 mg, single dose
  Arms: A
Drug: Doxazosin 4 mg ODT with water — Orally-disintegrating Tablet , 4 mg, single dose with water
  Arms: B
Drug: Doxazosin 4 mg ODT without water — Orally-disintegrating Tablet , 4 mg, single dose without water
  Arms: C

SUMMARY:
To test bioequivalence of Doxazosin 4 Mg Orally-disintegrating Tablet with Or Without Water to Doxazosin 4 Mg Japanese Marketed Immediate Release Tablet Under Fasted Condition

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy male subjects

Exclusion Criteria:

* Baseline orthostatic hypotension defined as a ≥20 mm Hg reduction in SBP, a ≥10 mm Hg reduction in DBP and/or the development of significant postural symptoms (dizziness, lightheadedness, vertigo) when going from the supine to standing position.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) and AUC from zero to the last sampling point (AUCt) of doxazosin 4 mg Orally Disintegrating Tablet (ODT) without water compared to doxazosin 4 mg Japanese marketed Immediate Release (IR) tablet under fasted conditions | up to 48 hours

SECONDARY OUTCOMES:
Cmax and AUCt of doxazosin 4 mg ODT with water compared to doxazosin 4 mg Japanese marketed IR tablet under fasted conditions. | up to 48 hours
Other Pharmacokinetic (PK) parameters (Tmax, AUC from zero to infinity (AUCinf), AUC from zero to the last measurable point (AUClast), elimination rate constant (Kel), t½, and mean residence time (MRT) of doxazosin under all forms of | up to 48 hours
administration. | up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0351069&StudyName=Bioequivalence%20Study%20of%20Doxazosin%204%20Mg%20Orally-Disintegrating%20Tablet%20With%20Or%20Without%20Water%20To%20Doxazosin%204%20Mg%20Japanese%20Marketed%20Immediate%20